CLINICAL TRIAL: NCT03514069
Title: Phase I Study of Ruxolitinib With Radiation and Temozolomide in Patients With Newly Diagnosed Grade III Gliomas and Glioblastoma
Brief Title: Ruxolitinib With Radiation and Temozolomide for Grade III Gliomas and Glioblastoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE3317
Record Dates: First submitted 2018-04-20; First posted 2018-05-02 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Glioma; Glioblastoma
Keywords: ruxolitinib; radiation; temozolomide
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — ruxolitinib; Radiation; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ruxolitinib + radiation x 60 Gy for 6 weeks (Experimental): Unmethylated O6-methylguanine DNA methyltransferase (MGMT) Glioblastoma and grade III glioma Every patient gets ruxolitinib + radiation x 60 Gy for 6 weeks over 6 weeks. The dose of radiation therapy is fixed at 60 Gy over 6 weeks
  Interventions: Drug: ruxolitinib; Radiation: radiation
- ruxolitinib + radiation x 60 Gy + temozolomide 75 mg/m (Experimental): Methylated MGMT Glioblastoma and grade III glioma. Arm 2 will start once the safe dose has been established for Arm 1 for every dose level.
  Every patient gets ruxolitinib + radiation x 60 Gy + daily temozolomide at 75 mg/m2 for 6 weeks over 6 weeks.
  The dose of radiation therapy is fixed at 60 Gy over 6 weeks (2 Gy x 30). The dose of temozolomide is 75 mg/m2 daily for 6 weeks
  Interventions: Drug: ruxolitinib; Radiation: radiation; Drug: temozolomide

INTERVENTIONS:
Drug: ruxolitinib — Starting dose ruxolitinib 10 mg twice daily
Radiation: radiation — 60gy for 6 weeks
Drug: temozolomide — 75mg/m2
  Arms: ruxolitinib + radiation x 60 Gy + temozolomide 75 mg/m

SUMMARY:
The purpose of this study is to test how well the drug works, safety and tolerability of an investigational drug called Ruxolitinib in gliomas and glioblastomas, when combined with standard treatment for brain cancer, temozolomide and radiation.

Ruxolitinib is an experimental drug that works by targeting proteins in cells and stops them from growing. Ruxolitinib is experimental because it is not approved by the Food and Drug Administration (FDA) for the treatment of gliomas or glioblastomas

Temozolomide works by damaging the DNA of tumor cells so that they cannot divide properly. Some tumor cells can repair that damage and therefore be resistant to temozolomide.

DETAILED DESCRIPTION:
Primary Objective

Arm 1:

To determine Maximum tolerated dose (MTD) of ruxolitinib with radiation (2 Gy x 30) in patients with unmethylated MGMT high-grade glioma (HGG)

Arm 2:

To determine Maximum tolerated dose (MTD) of ruxolitinib with radiation (2 Gy x 30) and daily temozolomide at 75 mg/m2 in patients with methylated MGMT high-grade glioma (HGG)

Secondary Objective(s)

Arm 1:

* Safety of combination of ruxolitinib with radiation
* Progression free survival (PFS)
* Overall survival (OS)

Arm 2:

* Safety of combination of ruxolitinib with radiation and temozolomide
* Progression free survival (PFS)
* Overall survival (OS)

STUDY DESIGN

A phase 1 design will be used with cohorts of 3 patients treated at each dose level in both arms 1 and 2 and monitored for treatment-related toxicities. Escalation to the next dose will proceed in the absence of dose-limiting toxicities (DLTs).

ELIGIBILITY:
Inclusion Criteria:

Arm 1:

* Patients must have unmethylated MGMT supratentorial high-grade glioma (anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic mixed astro oligodendroglioma or glioblastoma).

Arm 2:

* Patients must have supratentorial methylated MGMT high-grade glioma (anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic mixed astro oligodendroglioma or glioblastoma).

Both:

* Patients must have MRI or CT with contrast within 28 days prior to starting treatment.
* Patients must have a Karnofsky performance status ≥ 70% (i.e. the patient must be able to care for himself/herself with occasional help from others).
* Patients must have adequate blood, kidney and liver function
* Patients must be able to provide written informed consent.
* Patients and their sexual partners must agree to avoid conception while on the study due to possible risks from experimental drugs. Women will need a negative pregnancy test to be on the study
* Patients may not have any other cancers except skin cancer and localized bladder, prostate, cervical, or breast cancer which were cured more than 3 years ago

Exclusion Criteria:

* Patients with other serious diseases
* Pregnant women
* Patients getting other cancer treatments
* Patients with other cancers except for localized skin cancer and localized bladder, prostate, cervical, or breast cancer which were cured more than 3 years ago
* Patients who have had repeat craniotomy for tumor therapy after receiving radiation therapy and temozolomide treatment.
* Patients who have previously received other treatments for their cancers
* Patient has previously taken ruxolitinib or is allergic to components of the study drug
* Use of blood thinners
* Human immunodeficiency virus (HIV) infection
* Active hepatitis B or C infection
* Heart diseases including abnormal electrocardiogram (EKG)
* Patients unwilling or unable to follow this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of ruxolitinib with radiation in study patients | Up to 6 weeks
Maximum tolerated dose (MTD) of ruxolitinib with radiation and daily Temozolomide in study patients | Up to 6 weeks

SECONDARY OUTCOMES:
Number of patient study specific adverse events as a measure of safety | Up to 8 weeks after beginning treatment
  Study specific adverse events are defined as any of the following events occurring during the first 8 weeks of treatment with ruxolitinib and while being given radiation/temozolomide: grade 3 or 4 low platelets, grade 4 low red blood cells, grade 4 low white blood cells lasting more than a week, fever, any non-blood related side effect of grade 3 or greater (excluding hair loss) despite treatment, grade 4 radiation-related skin changes, and any episode of noninfectious pneumonitis.
Number of patients who have experienced progression free survival as defined by the response assessment in neuro-oncology (RANO) criteria | Up to 6 weeks
Average time patients stayed alive on study | Up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Peereboom, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States